CLINICAL TRIAL: NCT05560581
Title: Digital Self-efficacy Training to Bridge Waiting Times for Psychotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric University Hospital, Zurich (Other)
Responsible Party: Principal Investigator, Judith Rohde, MD, Clinician Scientist, Psychiatric University Hospital, Zurich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: SeApp III
Record Dates: First submitted 2022-09-25; First posted 2022-09-29 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-11

CONDITIONS: Psychiatric Disorder; Waiting for Psychotherapy
MeSH Terms: conditions — Mental Disorders | interventions — Ecological Momentary Assessment

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Participants will receive an one-week digital self-efficacy training (3x/day) and an one-week Ecological Momentary Assessment (3x/day questions on mood, social and virtual contacts).
  Interventions: Behavioral: Digital self-efficacy training; Behavioral: Ecological Momentary Assessment
- Control group (Active Comparator): Participants will receive an one-week Ecological Momentary Assessment (3x/day questions on mood, social and virtual contacts).
  Interventions: Behavioral: Ecological Momentary Assessment

INTERVENTIONS:
Behavioral: Digital self-efficacy training — Prior to the app participation, participants will receive psychoeducation on self-efficacy and will be instructed to define two autobiographical self-efficacy memories (own achievements, e.g., completion of an exam, success in a sporting event). During the week of app participation, they will be prompted three times per day and asked to perform an imagination task. Step by step, they will recall one of their autobiographic self-efficacy memories and focus on their character traits and abilities that were relevant for their achievement.
  Arms: Intervention group
Behavioral: Ecological Momentary Assessment — Participants will receive questions on mood and social/virtual contacts 3 times per day.

SUMMARY:
The main aim of this project is to improve waiting periods for specialised psychotherapy. We will apply a brief, smartphone-based self-efficacy training to patients with psychiatric disorders waiting for specialised psychotherapy. Additionally, we will use Ecological Momentary Assessment (EMA) to assess mood, social contacts, and other parameters daily. We will investigate whether the training can improve self-efficacy and related constructs and if it can help reduce stress and waitlist drop-outs during waiting periods. Additionally, we will investigate if the self-efficacy training has a positive effect on motivation and therapeutical relationship regarding the subsequent therapy.

After a screening for eligibility, participants will be randomly assigned to intervention and control group. At baseline, participants attend a laboratory session where they are assessed for current psychiatric disorders and further relevant psychological variables. They will then either participate in the digital self-efficacy training combined with EMA (intervention group) or in EMA only (control group). Both will be conducted via a smartphone app. Subsequently, participants will be asked to fill in post questionnaires at three different time points: after having finished app usage, one month later, and after the beginning of the subsequent psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* psychiatric disorder
* age 18-65
* waiting for psychiatric assessment/treatment (being on waitlist)
* sufficient knowledge of the German language
* smartphone user
* internet access via smartphone
* internet access at home (laptop, tablet, or computer)

Exclusion Criteria:

* current intense psychotherapy
* acute suicidality
* acute psychotic symptoms
* substance addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in self-efficacy | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Validated measures ("General Self-Efficacy Scale" (10 items; higher scores indicate higher self-efficacy -> better outcome), "Coping Self-efficacy scale" (26 items; higher scores indicate higher self-effiacy -> better outcome) and individual questions based on validated measures assessing specific self-efficacy regarding emotion regulation, therapy and waitlist will be used to assess self-efficacy at baseline and 3 different time points after the intervention.

SECONDARY OUTCOMES:
Change in hopelessness | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Hopelessness will be assessed using the validated measure "Beck Hopelessness Scale" (20 items; higher scores indicate greater hopelessness -> worse outcome).
Change in anxiety | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Anxiety will be assessed using the validated measure "State and Trait Anxiety Scale" (40 items; higher scores indicate greater anxiety -> worse outcome).
Change in stress | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Stress will be assessed using the validated measure "Perceived Stress Scale" (10 items; higher scores indicate greater stress -> worse outcome).
Change in therapy expectations | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Therapy expectations will be assessed using the validated measure "Patient Questionnaire on Therapy Expectation and Evaluation" (11 items; higher score indicates higher satisfaction -> better outcome).
Change in depression | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Depression will be assessed using the validated measure "Beck Depression Inventory II" (21 items; higher scores indicate greater depression -> worse outcome).
Change in optimism | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Change in life orientation will be assessed using the validated measure "Life Orientation Test Revised" (10 items; higher scores indicate greater optimism -> better outcome)
Change in intolerance of uncertainty | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Intolerance of uncertainty will be assessed using the validated measure "Intolerance of uncertainty scale" (18 items; higher scores indicate greater uncertainty -> worse outcome).

OTHER OUTCOMES:
Change in mood and contacts | 3 per day during one-week
  pos. and neg. mood and contacts will be assessed with the Ecological Momentary Assessment. Higher pos. mood / lower neg. mood -> better outcome
Change in in ability to work | baseline to 1 month after the intervention, within 1 month after the subsequent therapy began
  We will ask about the participants' self-evaluation at baseline and 2 different time points after the intervention (self-evaluation; no specific score will be used)
Motivation and life enjoyment | baseline to 1 day after the intervention, 1 month after the intervention, within 1 month after the subsequent therapy began
  Additional questionnaire with single items assessing therapy motivation and life enjoyment with items based on the validated questionnaires "Quality of Life Enjoymend and Satisfaction Questionnaire", "Fragebogen zur Psychotherapiemotivation" und "Fragebogen zur Messung der Psychotherapiemotivation"

CONTACTS AND LOCATIONS:
Overall Officials: Judith Rohde, MD, Principal Investigator — Psychiatric University Hospital Zurich, University of Zurich
Locations (2):
- Switzerland (2):
  - Integrated Psychiatry Winterthur, Winterthur
  - Psychiatric University Hospital, Zurich

IPD SHARING:
Plan to Share IPD: Undecided